CLINICAL TRIAL: NCT01200810
Title: A Randomized Phase II Study of Peripheral Androgen Blockade With Bicalutamide Followed by Placebo or Treatment With the Gamma Secretase Inhibitor RO4929097 in Men With Rising PSA After Definitive Local Therapy for Adenocarcinoma of the Prostate
Brief Title: Bicalutamide and RO4929097 in Treating Patients With Previously Treated Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug was no longer available
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-02527; CINJ-081001 (Other: CINJ); CDR0000684276 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; bicalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Placebo Comparator): Patients receive oral placebo once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Drug: bicalutamide
- Arm II (Experimental): Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Drug: bicalutamide

INTERVENTIONS:
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm I
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Drug: bicalutamide — Given orally
  Other Names: Casodex; CDX

SUMMARY:
This partially randomized phase II trial is studying how well giving bicalutamide together with RO4929097 works in treating patients with previously treated prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, may lessen the amount of androgens made by the body. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bicalutamide together with RO4929097 may be an effective treatment for prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the difference in the time to PSA progression in patients with adenocarcinoma of the prostate who have rising PSA after definitive local therapy treated with bicalutamide with vs without gamma-secretase/Notch signalling pathway inhibitor RO4929097 (RO4929097).

SECONDARY OBJECTIVES:

I. To determine the proportion of patients from each arm who achieve complete response (by PSA) during the combination phase.

II. To determine the proportion of patients from each arm with PSA progression during the combination phase.

III. To determine the time to PSA nadir during the combination phase for patients in each arm.

IV. To determine the time to PSA progression during the combination phase for patients in each arm.

V. To determine the time to PSA progression during the observation phase. VI. To determine the proportion of patients with PSA progression during the observation phase.

VII. To assess the safety and tolerability of gamma-secretase inhibitor RO4929097 in combination with bicalutamide.

VIII. To evaluate expression for targets of gamma secretase inhibitor in a prostate tissue microarray.

IX. To collect serum for future evaluation of soluble markers of gamma-secretase inhibition and angiogenesis.

OUTLINE: This is a multicenter study.

INDUCTION PHASE: All patients receive induction therapy comprising oral bicalutamide once daily for at least 16 weeks. Patients whose PSA declines at least 50% continue to the randomization phase.

RANDOMIZATION PHASE: Patients are stratified according to prior therapy (radiotherapy vs surgery) and randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral placebo once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.

ARM II: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO4929097 (RO4929097) once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.

Patients with no disease progression continue to the combination phase. Patients with disease progression undergo imaging studies to verify the absence of metastatic disease before continuing to the combination phase.

COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples may be collected periodically for correlative studies. After completion of study treatment, patients are followed up every 6 weeks for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer

  * Stage D0 OR D1 disease (i.e., tumor originally diagnosed as being limited to the prostate and regional lymph nodes)
  * Has a rising PSA value after definitive local therapy (i.e., prostatectomy or radiotherapy) and no radiographic evidence of disease
* PSA progression after local treatment:

  * PSA values for patients after surgery must be ≥ 0.2 ng/mL, determined by two measurements, ≥ 1 month apart and ≥ 6 months after prostatectomy
  * PSA values for patients after radiotherapy must be ≥ 2.0 ng/mL above the nadir PSA achieved after radiotherapy, determined by two measurements at 1 month apart and ≥ 6 months after completion of the radiotherapy treatment (patients who received adjuvant or salvage radiotherapy after prostatectomy must have PSA of ≥ 0.2 ng/mL)
  * The first two PSA values, along with a third (study baseline) value must all be rising (i.e., there must be an overall rising trajectory, such that the third value cannot be lower than the first value)
* No metastatic disease on baseline bone scan and CT scan of the abdomen/pelvis
* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 40 mL/min for patients with creatinine levels above normal
* Bilirubin normal
* AST and/or ALT ≤ 2.5 times ULN
* Serum total testosterone level ≥ 150 ng/dL
* No uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia, defined as less than the lower limit of normal despite adequate electrolyte supplementation
* Fertile patients must use two effective forms of contraception (i.e., barrier contraception and one other method of contraception) for 1 week before, during, and for ≥ 12 months after completion of study treatment
* Able to swallow tablets
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * A history of torsades de pointes
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness or social situation that would limit compliance with study requirements
* Baseline QTc ≤ 450 msec
* No serologic positivity for acute hepatitis A, acute or chronic hepatitis B, or acute or chronic hepatitis C
* No history of liver disease or other forms of hepatitis or cirrhosis
* No HIV-positive patients on combination antiretroviral therapy
* No serious concurrent systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or bicalutamide
* Patients may not donate sperm or blood during or for ≥ 12 months after completion of study treatment
* No concurrent medications or food that may interfere with the metabolism of RO4929097 including grapefruit and fresh-squeezed grapefruit juice
* Recovered from adverse events to < CTCAE grade 2
* At least 3 months since prior and no concurrent androgen-deprivation therapy (ADT)

  * Hormone-ablative treatment is only allowed in the neoadjuvant setting or in the setting of primary or salvage radiotherapy
  * No more than 36 months of neoadjuvant/ adjuvant ADT
* More than 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior and no concurrent estrogens, estrogen-like substances (i.e., PC-SPES, saw palmetto, or other herbal product that may contain phytoestrogens), or any other hormonal therapy (including flutamide, nilutamide, finasteride, ketoconazole, systemic corticosteroids, megestrol acetate, or cyproterone acetate)
* No other concurrent investigational agents
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4
* No other investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy, including chemotherapy, immunotherapy, hormonal cancer therapy, radiotherapy, or surgery for cancer
* No concurrent hormonal therapy with a leuteinizing hormone-releasing hormone (LHRH) agonist therapy (e.g., leuprolide or goserelin) or LHRH antagonist (e.g., abarelix)
* No concurrent growth factors (e.g., G-CSF), packed RBC transfusions, or platelet transfusions
* No concurrent antiarrhythmics or other medications known to prolong QTc

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, Principal Investigator — UMDNJ - Robert Wood Johnson University Hospital
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 patients were enrolled from a comprehensive cancer center in central New Jersey from August 2010 through November 2011.
Pre-assignment Details: During the induction phase, if subjects do not have a decline in PSA ≥ 50%, they are taken off study. Subjects who have a PSA decline ≥ 50% are randomized to Arm I or Arm II.
Groups:
- Arm I - Placebo: Patients receive oral placebo once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given orally
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bicalutamide: Given orally
- Arm II - RO4929097: Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bicalutamide: Given orally
Period: Overall Study
Arm/Group | Arm I - Placebo | Arm II - RO4929097
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Sponsor stopped making study drug | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive oral placebo once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given orally
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bicalutamide: Given orally
- Arm II: Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Treatment repeats every 21 days for 18 courses in the absence of PSA progression.
  COMBINATION PHASE: All patients then receive oral bicalutamide once daily on days 1-21 and oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bicalutamide: Given orally
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (6.28) | 67.6 (7.5) | 64.8 (7.16)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to PSA Progression
Description: Time to PSA progression will be compared in the two groups using a log-rank test for a maximum of 54 weeks.
Time Frame: Up to 12 months
Population: Data were not collected as the protocol was terminated early due to lack of study drug. Only three patients progressed during randomization phase.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Patients Who Achieve Complete Response (by PSA) During the Combination Phase
Time Frame: Up to 12 months
Population: Data were not collected as study was terminated early due to lack of study drug. Only three patients started combination phase and were then removed from study due to lack of study drug.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Patients With PSA Progression During the Combination Phase
Time Frame: Up to 12 months
Population: as for outcome 2
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to PSA Nadir During the Combination Phase
Time Frame: Up to 12 months
Population: Data were not collected as study was terminated early due to lack of study drug.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to PSA Progression During the Combination Phase
Time Frame: Up to 12 months
Population: Data were not collected as study was terminated early due to lack of study drug.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to PSA Progression During the Observation Phase
Time Frame: Up to 12 months
Population: Data were not collected as study was terminated early due to lack of study drug. No subjects entered the observation phase.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Proportion of Patients With PSA Progression During the Observation Phase
Time Frame: Up to 12 months
Population: as for outcome 6
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Safety and Tolerability Assessed Using NCI CTCAE Version 4.0
Description: Number of participants randomized to RO4929097 arm who experienced serious adverse events .
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm I - Placebo | Arm II - RO4929097
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Placebo (N=5) | Arm II - RO4929097 (N=5)
Hyphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
lightheadedness (Nervous system disorders) | 0 | 1 (1)
hot flashes (Vascular disorders) | 0 (0) | 2 (3)
constipation with blood (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (2)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthritic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral eye infection (Infections and infestations) | 0 (0) | 1 (1)
Contact dermatitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased lymphocytes (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Elevated Alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
Elevated ALT (Investigations) | 0 (0) | 1 (1)
Erythematous right shin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythematous rash (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Low phosphorous (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
leukopenia (Investigations) | 1 (1) | 0 (0)
lymphopenia (Investigations) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritic macular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rhinorrhea (Infections and infestations) | 0 (0) | 1 (1)
Right fore arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less